CLINICAL TRIAL: NCT04131322
Title: Loss of Response of Adalimumab Biosimilar Compared With the Loss of Response of Adalimumab Original: Controlled, Randomized, Non-inferiority Open Study. "ADA-SWITCH Study"
Brief Title: Loss of Response of Adalimumab Biosimilar vs Adalimumab Original, in Inflammatory Bowel Disease.
Acronym: ADA-SWITCH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor cancellation
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMGEVITA-HVM2019
Record Dates: First submitted 2019-10-10; First posted 2019-10-18 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Crohn Disease; Ulcerative Colitis
Keywords: Loss of response; Switching; Adalimumab original; Adalimumab biosimilar
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Solutions; Injections; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- switch-cohort (Experimental): Adalimumab biosimilar
  Interventions: Drug: Amgevita 40Mg Solution for Injection
- non-switchcohort (Active Comparator): Adalimumab original
  Interventions: Drug: HUMIRA 40Mg Solution for Injection

INTERVENTIONS:
Drug: Amgevita 40Mg Solution for Injection — Adalimumab 40Mg Solution for Injection
  Other Names: AMGEVITA
  Arms: switch-cohort
Drug: HUMIRA 40Mg Solution for Injection — Adalimumab 40Mg Solution for Injection
  Other Names: HUMIRA
  Arms: non-switchcohort

SUMMARY:
Loss of response of the Adalimumab biosimilar compared with the original drug.

DETAILED DESCRIPTION:
A single-site Unicentric, randomized, parallel-group, non-inferiority open study including patients diagnosed with inflammatory bowel disease (Crohn's disease and Ulcerative Colitis) who were in clinical remission with Adalimumab original for at least 6 months prior to the start of the study.

A total of 216 patients with inflammatory bowel disease from the Inflammatory Unit of the Virgin Macarena University Hospital will be randomized 1:1 to receive the study drug, Adalimumab biosimilar (AMGEVITA®) subcutaneous 40mg every 15 days or maintain the original drug (Humira®) 40 mg subcutaneous every 15 days.

The dosage of the medication will be administrated according to the product's approved label by SmPC (Summary of Product's Characteristics)by technical file. Administration will be accepted every 7 days, if the patient after inclusion criteria is included with intensified dose.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female over 18 years of age
* Be a Patient with a previous confirmed diagnosis of Crohn´s disease an Ulcerative Colitis
* Previous treated with original Adalimumab for at least 6 months with regular maintenance dose (40 mg every 15 days) and in clinical and biological remission.
* Patients under treatment with intensified Adalimumab (40mg every 7 days or 80mg every 7 days) to maintain clinical and biological remission for at least 6 months.
* Patients with oral mesalazine with a stable dose for more than 30 days.
* Patients with immunosuppressive therapy (methotrexate, azathioprine) with a minimum intake time> 60 days.
* Patients may be accepted with corticosteroids at the established doses:

prednisone <20mg / dl, budesonide <9mg / dl.

* Patients who have a tuberculosis (TB) study (Mantoux / QuantiFERONTB test) updated in the last two year, with a negative result.
* Patient with serology hepatitis B and C, updated at the beginning of the treatment with Humira®
* Sign an informed consent document indicating that he/she understands the purpose of, and procedures required for, the study and are willing to participate in the study.

Exclusion Criteria:

* Positive pregnancy test at the time of inclusion or during the follow-up period, as well as women who are breastfeeding
* Patients with uncontrolled comorbidities, active cancer, diabetes mellitus, severe cardiovascular disease, obstructive pulmonary disease, serious active infections.
* Patients with oral mesalazine initiated less than 30 days.
* Patients with immunosuppressive therapy (methotrexate, azathioprine) with a minimum intake time of <60 days.
* Patient with original Adalimumab who do not meet a minimum of 6 months of stable dose (40 mg every 7 or 15 days)
* Patient on corticosteroid therapy at doses: prednisone> 20mg / dl, budesonide = 9mg / dl, or with IV corticoids within 14 days prior screening date.
* Patients with mental disorders, alcohol / other substance abuse, or conditions that do not allow adherence to the study protocol.
* Patients with active TB
* Patients with defined Hepatitis B and C defined as:

HBV: hepatitis B surface antigen (HbsAg) positive together with positive HBV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR). HCV: HCV ribonucleic acid (RNA) detectable in any patient with positive anti-HCV antibody (IgG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline to final follow-up in the response of the switch. | From date of randomization until the date of first documented change from baseline status in concomitant steroids needed or increment in dose or frequency of adalimumab biosimilar or urgent surgery indication ever came first, assessed up to 13 months
  To assess if there is a change in the response of the switch (replacement) from Adalimumab original (Humira®) to Adalimumab biosimilar (Amgevita®) trhough the quantification of concomitant steroids needed or increment in dose or frequency of adalimumab biosimilar or urgent surgery indication

SECONDARY OUTCOMES:
Compare the antibody formation rate. | 0, 3, 6, 9, 12, 13 months
  Compare the antibody formation rate with Adalimumab(immunogenicity) after the switch.
The score of the specific quality of life questionnaire | 0, 3, 6, 9, 12, 13 months
  Compare the score of the specific quality of life questionnaire Short Inflammatory Bowel Disease Questionnaire (SIBDQ) in patients with inflammatory bowel disease before and after the switch.The minimum value is 1 and the maximum is 7, where higher scores means better outcome.
The score of the Visual Analogue Scale (VAS) | 0, 3, 6, 9, 12, 13 months
  Compare the score of the Visual Analogue Scale (VAS) of pain at the puncture site after the switch. The minimum value is 0 mm and the maximum value is 100 mm, where the higher score means a worse outcome.
Maintenance of bioquimical remission trhough C-reactive protein | 0, 3, 6, 9, 12, 13 months
  levels of C-reactive protein in blood (mg/L).
Maintenance of bioquimical remission through Calprotectin values | 0, 3, 6, 9, 12, 13 months
  levels of Calprotectin in blood (µg/g).
Drug levels | 0, 3, 6, 9, 12, 13 months
  Determination of drug levels in blood (µg/ml).
Adverse Event | 0, 3, 6, 9, 12, 13 months
  Proportion of patients who experience AE in each treatment group
Hospital admission rate | 0, 3, 6, 9, 12, 13 months
  Proportion of patients requiring hospital admissions related to a disease outbreak during follow-up.
Surgery rate | 0, 3, 6, 9, 12, 13 months
  Proportion of patients requiring surgery related to disease activity during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Argüelles Arias, Md PhD, Principal Investigator — Universitary Hospital Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: No